CLINICAL TRIAL: NCT03458559
Title: Repeated Rhenium-188-HEDP Versus Radium-223-chloride in Patients With Metastatic Castration-resistant Prostate Cancer: The RaRe Study
Brief Title: Rhenium-188-HEDP vs. Radium-223-chloride in Patients With Advanced Prostate Cancer Refractory to Hormonal Therapy
Acronym: RaRe
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, A.J.M. van den Eertwegh, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017.610
Record Dates: First submitted 2018-02-14; First posted 2018-03-08 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer Metastatic to Bone
Keywords: Bone metastases; Rhenium-188-HEDP; Radium 223-chloride; Survival; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride; rhenium-186 HEDP

STUDY DESIGN:
Intervention Model Description: Patients will be randomized between
  * radium-223-chloride intravenously, for a total of 6 administrations (every 4weeks)
  * rhenium-188-HEDP intravenously for a total of 3 administratrions (every 8 weeks)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radium-223-chloride (Active Comparator): Radium-223-chloride 50kBg/kg, every 4 weeks intravenously, for a total of 6 administrations.
  Interventions: Drug: Radium-223 chloride
- Rhenium-188-HEDP (Experimental): Rhenium-188-HEDP 40MBq/kg, every 8 weeks intravenously, for a total of 3 administrations.
  Interventions: Drug: Rhenium-188-HEDP

INTERVENTIONS:
Drug: Radium-223 chloride — Intravenously 50 kBq/kg every 4 weeks. Total: 6 administrations
  Other Names: Xofigo; Radium-223 dichloride
  Arms: Radium-223-chloride
Drug: Rhenium-188-HEDP — Intravenously 40 MBq/kg every 8 weeks. Total: 3 administrations
  Other Names: Re-188-HEDP; 188Rhenium-etidronate
  Arms: Rhenium-188-HEDP

SUMMARY:
Radium-223 chloride is an alpha-emitting radiopharmaceutical with proven survival benefit in patients with castration-resistant prostate cancer metastatic to bone. Beta-emitting radiopharmaceuticals have proven efficacy for palliating malignant bone pain. Nowadays, rhenium-188-HEDP is used in clinical practice for pain relief and palliative care. Several studies suggest that also rhenium-188-HEDP has the potential to improve overall survival. The purpose of this study is to investigate if treatment with rhenium-188-HEDP results in improvement of overall survival compared to treatment with radium-223-chloride.

DETAILED DESCRIPTION:
The main objective of this trial is to compare rhenium-188-HEDP (a beta-emitting radiopharmaceutical) with radium-223-chloride (an alfa-emitting radiopharmaceutical), in patients with castration-resistant prostate cancer metastatic to bone, with overall survival as primary endpoint.

For radium-223-chloride, an overall survival benefit has been proven in a large randomized phase III trial. Although such a trial has never been performed for rhenium-188-HEDP, some trials in literature suggest a survival benefit for rhenium as well.

Rhenium has some advantages compared to radium. Firstly, it is easily available as it can be produced in the hospital. Secondly, the costs of rhenium are significantly lower compared to radium. Lastly, rhenium seems to have a favorable pain response. However, no randomized trials have been performed to confirm this.

ELIGIBILITY:
Inclusion Criteria:

* Male, 18 years or older
* Histologically confirmed prostate cancer
* Bone metastases (≥ 6 lesions) showing pathological uptake at bone scintigraphy.
* WHO performance status of ≤2
* Life expectancy of at least 6 months
* Castration-resistant disease: serum testosterone level of ≤ 1.7 nmol per liter (≤50 ng per deciliter) after bilateral orchiectomy or during maintenance treatment consisting of androgen-ablation therapy with a luteinizing hormone-releasing hormone agonist. During study treatment the maintenance androgen-deprivation therapy must be continued.
* Baseline PSA ≥5 ng/ml with evidence of progressively increasing PSA values
* Symptomatic disease with either regular use of analgesic medication or treatment with external-beam radiotherapy for cancer-related bone pain within the previous 12 weeks.
* Progression on or after treatment with docetaxel, or inability to receive docetaxel.
* Adequate renal function (serum creatinine level ≤1.5 x ULN)
* Adequate hematological function defined as absolute neutrophil count ≥ 1.5x10^9/L and platelet count ≥100x 10^9/L)
* Written informed consent

Exclusion Criteria:

* Treatment with chemotherapy within the previous 4 weeks
* Continuation of treatment with abiraterone or enzalutamide
* Previous hemibody external radiotherapy
* Systemic radiotherapy with radioisotopes within the previous 24 weeks
* Malignant lymphadenopathy ≥3cm in the short-axis diameter
* Presence of visceral metastases
* Imminent of established spinal cord compression
* Active uncontrolled bacterial, viral or fungal infection
* History of another malignancy within the last five years except adequately treated basal cell carcinoma of the skin
* Organ allografts requiring immunosuppressive therapy.
* Any serious uncontrolled concommitant disease
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule: those conditions should be discussed with the patient before registration in the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2018-05-16 (Actual); Primary Completion 2022-05-16 (Estimated); Study Completion 2024-05-16 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Time from randomization until death due to any cause, an average of 18 months
  Time from randomization until death due to any cause,

SECONDARY OUTCOMES:
Time to PSA progression | Time from randomization to the date of a minimum of rising PSA levels, an average of 8 months (PSA measured at baseline and every 4 weeks).
  Time from randomization to the date of a minimum of rising PSA levels with an interval of >1week between each determination
Time to total-ALP progression | Time from randomization to the date of earliest objective evidence of ALP progression, an average of 8 months (ALP measure at baseline and every 4 weeks)
  Time from randomization to the date of earliest objective evidence of ALP progression.
Clinical progression | Time from randomization to the date of first clinical progression, an average of 12 months
  Time from randomization to the date of first clinical progression.
Time to first SRE | Time from randomization to the date of first skeletal related events, an average of 12 months
  Time from randomization to the date of first skeletal related events
Quality of life | Assessed through study completion, an average of 1 year
  Measured by the EORTC quality of Life Questionnaire C30
Effect on pain | Assessed through study completion, an average of 1 year
  Measured with a visual analogue scale
Incremental Cost Effectiveness Ratio (IVER) | Assessed through study completion, an average of 1 year
  Ratio between the difference in costs and the difference in benefits (quality of life of treatment with rhenium-188-HEDP of radium-223-chloride)

CONTACTS AND LOCATIONS:
Overall Officials: Alfons JM van den Eertwegh, Prof.dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palmedo H, Manka-Waluch A, Albers P, Schmidt-Wolf IG, Reinhardt M, Ezziddin S, Joe A, Roedel R, Fimmers R, Knapp FF Jr, Guhlke S, Biersack HJ. Repeated bone-targeted therapy for hormone-refractory prostate carcinoma: tandomized phase II trial with the new, high-energy radiopharmaceutical rhenium-188 hydroxyethylidenediphosphonate. J Clin Oncol. 2003 Aug 1;21(15):2869-75. doi: 10.1200/JCO.2003.12.060. PMID 12885803
- [Background] Biersack HJ, Palmedo H, Andris A, Rogenhofer S, Knapp FF, Guhlke S, Ezziddin S, Bucerius J, von Mallek D. Palliation and survival after repeated (188)Re-HEDP therapy of hormone-refractory bone metastases of prostate cancer: a retrospective analysis. J Nucl Med. 2011 Nov;52(11):1721-6. doi: 10.2967/jnumed.111.093674. Epub 2011 Oct 5. PMID 21976530
- [Background] Jong JM, Oprea-Lager DE, Hooft L, de Klerk JM, Bloemendal HJ, Verheul HM, Hoekstra OS, van den Eertwegh AJ. Radiopharmaceuticals for Palliation of Bone Pain in Patients with Castration-resistant Prostate Cancer Metastatic to Bone: A Systematic Review. Eur Urol. 2016 Sep;70(3):416-26. doi: 10.1016/j.eururo.2015.09.005. Epub 2015 Sep 19. PMID 26391636